CLINICAL TRIAL: NCT01953276
Title: Are Serial Electrocardiograms Additive to SeriAl Second-generations Troponins in Predicting Acute CoronAry Syndromes in PatienTs With Undifferentiated cHest Pain (ASAP CATH) Study
Brief Title: Are Serial Electrocardiograms Additive to SeriAl Second-generations Troponins in Predicting Acute CoronAry Syndromes in PatienTs With Undifferentiated cHest Pain
Acronym: ASAP Cath
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00022288
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2018-02

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: Acute Coronary Syndrome; Chest pain; Electrocardiograms; Risk Stratification; Emergency Department
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples are obtained from patients and processed so that the plasma is extracted and frozen for future research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Serial Electrocardiogram Arm: All study participants will receive serial electrocardiograms.
  Interventions: Device: Serial Electrocardiograms

INTERVENTIONS:
Device: Serial Electrocardiograms — All participants will have serial electrocardiograms performed.

SUMMARY:
Our research will examine whether the presence or absence of serial electrocardiogram (ECG) changes aids in reclassifying participants' risk for major adverse cardiac events (MACE) over and above serial blood testing.

DETAILED DESCRIPTION:
Chest pain is one of the most common symptoms evaluated in the Emergency Department (ED). One of the primary diagnostic concerns during the evaluation of this presentation is whether there is evidence of acute coronary syndromes (ACS) as ACS is a major risk factor for short- and long-term major adverse cardiovascular events (MACE, defined as acute myocardial infarction, revascularization, or all-cause death). Two of the cornerstones of the guidelines-based evaluation of this patient group are serial electrocardiograms (ECG) and troponin measurements (a serological marker of myocardial ischemia), which have shown to be both independently and incrementally predictive of ACS. Recently, second-generation troponin assays have been adopted into clinical practice as they have higher sensitivity and specificity for ACS compared to older assays. Given the increased diagnostic accuracy of these novel second-generation assays, the proposed study's research question is to investigate whether serial ECG changes significantly increase the diagnostic accuracy of serial second-generation troponin changes in predicting MACE in patients presenting with symptoms consistent with ACS. In order to investigate this question, we originally proposed an observational pilot study ancillary to the HEART Pathway trial (WFUHS IRB00021074), a funded randomized controlled trial investigating a recently developed decision aid tool (the HEART score) designed to identify patients being evaluated for chest pain that can safely forgo further objective testing. We proposed to add the collection of two additional 12-lead ECGs to the protocol in the HEART Pathway trial, which included serial second-generation troponin collection, in order to generate pilot data regarding the research question. As recruitment for the HEART Pathway trial ended in February 2014, we now propose to continue enrollment for the ASAP CATH study independently, as a prospective observational study evaluating the additional prognostic value of serial ECGs to standard care in patients with chest pain being evaluated for acute coronary syndromes in the Emergency Department.

Objective:

The goal of this project is to produce preliminary data to investigate whether the presence or absence of serial ECG changes suggestive of myocardial ischemia aids in reclassifying participants' risk for MACE and objective evidence of ACS over and above serial second-generation troponin testing.

Methods:

Adult patients, over 21 years old, presenting to WFBMC ED with chest pain or symptoms concerning for ACS, in which the provider orders cardiac biomarkers and an ECG will be eligible for enrollment. We aim to add serial ECG analysis (one at the time of study enrollment and a second at the time of the study blood draw) to the protocol in the proposed study. The primary outcomes are major adverse cardiovascular events (MACE) at 30 days and evidence of acute myocardial ischemia via objective cardiac testing performed during the index hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 21 years of age at the time of enrollment
* Chest discomfort or other symptoms consistent with possible ACS as indicated by the treating physician after obtaining an ECG and cardiac biomarkers for the patient's evaluation
* The treating physician feels the patient could be discharged home if cardiac disease was excluded

Exclusion Criteria:

* Evidence of ST-elevation myocardial infarction (STEMI) or left bundle branch block (LBBB) on initial ECG
* Left ventricular systolic dysfunction (history of left ventricular ejection fraction <40% or active symptoms of congestive heart failure)
* New or uncontrolled ventricular arrhythmias on initial ECG
* Hemodynamic instability: heart rate > 120 bpm or < 40 bpm and/or systolic blood pressure <100 mmHg
* Hypoxemia (oxygen saturation <90% on room air or normal home oxygen flow rate)
* Terminal diagnosis with life expectancy less than 1 year
* A non-cardiac medical, surgical, or psychiatric illness determined by the provider to require admission, increase risk of objective cardiac testing, or prevent immediate discharge following negative testing.
* Prior enrollment
* Incapacity or unwillingness to provide consent and comply with study procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Wake Forest Baptist Health Emergency Department with symptoms concerning for Acute Coronary Syndrome (ACS) are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events at 30 days | 30 Days
  Determine whether serial electrocardiogram changes significantly increase the diagnostic accuracy of serial second-generation troponin measurements in predicting MACE at 30 days in patients with symptoms suggestive of ACS.
Evidence of acute myocardial ischemia via objective cardiac testing performed during the index hospitalization | Duration of initial hospitalization, usually 1 to 2 days
  Determine whether serial ECG changes significantly increase the diagnostic accuracy of serial second-generation troponin measurements in predicting positive cardiac stress testing or coronary angiography findings indicative of acute myocardial ischemia in patients being evaluated for ACS.
Major Adverse Cardiovascular Events at 30 days | 30 Days
  Determine whether serial ECG changes significantly increase the diagnostic accuracy of serial second-generation troponin measurements in predicting major adverse cardiovascular events at 30 days in patients with symptoms suggestive of ACS.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mahler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center - Emergency Department, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Owens PL, Barrett ML, Gibson TB, Andrews RM, Weinick RM, Mutter RL. Emergency department care in the United States: a profile of national data sources. Ann Emerg Med. 2010 Aug;56(2):150-65. doi: 10.1016/j.annemergmed.2009.11.022. Epub 2010 Jan 15. PMID 20074834
- [Background] Mahler SA, Hiestand BC, Goff DC Jr, Hoekstra JW, Miller CD. Can the HEART score safely reduce stress testing and cardiac imaging in patients at low risk for major adverse cardiac events? Crit Pathw Cardiol. 2011 Sep;10(3):128-33. doi: 10.1097/HPC.0b013e3182315a85. PMID 21989033
- [Background] Hedges JR, Young GP, Henkel GF, Gibler WB, Green TR, Swanson JR. Serial ECGs are less accurate than serial CK-MB results for emergency department diagnosis of myocardial infarction. Ann Emerg Med. 1992 Dec;21(12):1445-50. doi: 10.1016/s0196-0644(05)80057-5. PMID 1443839
- [Background] Fesmire FM, Percy RF, Bardoner JB, Wharton DR, Calhoun FB. Usefulness of automated serial 12-lead ECG monitoring during the initial emergency department evaluation of patients with chest pain. Ann Emerg Med. 1998 Jan;31(1):3-11. doi: 10.1016/s0196-0644(98)70274-4. PMID 9437335
- [Background] Carmo P, Ferreira J, Aguiar C, Ferreira A, Raposo L, Goncalves P, Brito J, Silva A. Does continuous ST-segment monitoring add prognostic information to the TIMI, PURSUIT, and GRACE risk scores? Ann Noninvasive Electrocardiol. 2011 Jul;16(3):239-49. doi: 10.1111/j.1542-474X.2011.00438.x. PMID 21762251
- [Background] Yan AT, Yan RT, Tan M, Senaratne M, Fitchett DH, Langer A, Goodman SG; INTERACT Investigators. Long-term prognostic value and therapeutic implications of continuous ST-segment monitoring in acute coronary syndrome. Am Heart J. 2007 Apr;153(4):500-6. doi: 10.1016/j.ahj.2007.02.003. PMID 17383285
- [Background] Jernberg T, Lindahl B, Wallentin L. The combination of a continuous 12-lead ECG and troponin T; a valuable tool for risk stratification during the first 6 hours in patients with chest pain and a non-diagnostic ECG. Eur Heart J. 2000 Sep;21(17):1464-72. doi: 10.1053/euhj.2000.2178. PMID 10952839
- [Background] Norgaard BL, Andersen K, Dellborg M, Abrahamsson P, Ravkilde J, Thygesen K. Admission risk assessment by cardiac troponin T in unstable coronary artery disease: additional prognostic information from continuous ST segment monitoring. TRIM study group. Thrombin Inhibition in Myocardial Ischemia. J Am Coll Cardiol. 1999 May;33(6):1519-27. doi: 10.1016/s0735-1097(99)00080-7. PMID 10334417
- [Background] Fesmire FM, Decker WW, Diercks DB, Ghaemmaghami CA, Nazarian D, Brady WJ, Hahn S, Jagoda AS; American College of Emergency Physicians Clinical Policies Subcommittee (Writing Committee) on Non-ST-Segment Elevation Acute Coronary Syndromes. Clinical policy: critical issues in the evaluation and management of adult patients with non-ST-segment elevation acute coronary syndromes. Ann Emerg Med. 2006 Sep;48(3):270-301. doi: 10.1016/j.annemergmed.2006.07.005. No abstract available. PMID 16934648
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr; 2011 WRITING GROUP MEMBERS; ACCF/AHA TASK FORCE MEMBERS. 2011 ACCF/AHA Focused Update Incorporated Into the ACC/AHA 2007 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 May 10;123(18):e426-579. doi: 10.1161/CIR.0b013e318212bb8b. Epub 2011 Mar 28. No abstract available. PMID 21444888
- [Background] Antman EM, Tanasijevic MJ, Thompson B, Schactman M, McCabe CH, Cannon CP, Fischer GA, Fung AY, Thompson C, Wybenga D, Braunwald E. Cardiac-specific troponin I levels to predict the risk of mortality in patients with acute coronary syndromes. N Engl J Med. 1996 Oct 31;335(18):1342-9. doi: 10.1056/NEJM199610313351802. PMID 8857017
- [Background] Alpert JS, Thygesen K, Antman E, Bassand JP. Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. J Am Coll Cardiol. 2000 Sep;36(3):959-69. doi: 10.1016/s0735-1097(00)00804-4. PMID 10987628
- [Background] Luepker RV, Apple FS, Christenson RH, Crow RS, Fortmann SP, Goff D, Goldberg RJ, Hand MM, Jaffe AS, Julian DG, Levy D, Manolio T, Mendis S, Mensah G, Pajak A, Prineas RJ, Reddy KS, Roger VL, Rosamond WD, Shahar E, Sharrett AR, Sorlie P, Tunstall-Pedoe H; AHA Council on Epidemiology and Prevention; AHA Statistics Committee; World Heart Federation Council on Epidemiology and Prevention; European Society of Cardiology Working Group on Epidemiology and Prevention; Centers for Disease Control and Prevention; National Heart, Lung, and Blood Institute. Case definitions for acute coronary heart disease in epidemiology and clinical research studies: a statement from the AHA Council on Epidemiology and Prevention; AHA Statistics Committee; World Heart Federation Council on Epidemiology and Prevention; the European Society of Cardiology Working Group on Epidemiology and Prevention; Centers for Disease Control and Prevention; and the National Heart, Lung, and Blood Institute. Circulation. 2003 Nov 18;108(20):2543-9. doi: 10.1161/01.CIR.0000100560.46946.EA. Epub 2003 Nov 10. No abstract available. PMID 14610011
- [Background] Norgaard BL, Andersen K, Thygesen K, Ravkilde J, Abrahamsson P, Grip L, Dellborg M. Long term risk stratification of patients with acute coronary syndromes: characteristics of troponin T testing and continuous ST segment monitoring. Heart. 2004 Jul;90(7):739-44. doi: 10.1136/hrt.2003.020479. PMID 15201240
- [Background] Keller T, Zeller T, Peetz D, Tzikas S, Roth A, Czyz E, Bickel C, Baldus S, Warnholtz A, Frohlich M, Sinning CR, Eleftheriadis MS, Wild PS, Schnabel RB, Lubos E, Jachmann N, Genth-Zotz S, Post F, Nicaud V, Tiret L, Lackner KJ, Munzel TF, Blankenberg S. Sensitive troponin I assay in early diagnosis of acute myocardial infarction. N Engl J Med. 2009 Aug 27;361(9):868-77. doi: 10.1056/NEJMoa0903515. PMID 19710485
- [Background] Katus HA, Remppis A, Neumann FJ, Scheffold T, Diederich KW, Vinar G, Noe A, Matern G, Kuebler W. Diagnostic efficiency of troponin T measurements in acute myocardial infarction. Circulation. 1991 Mar;83(3):902-12. doi: 10.1161/01.cir.83.3.902. PMID 1999039
- [Background] Melanson SE, Morrow DA, Jarolim P. Earlier detection of myocardial injury in a preliminary evaluation using a new troponin I assay with improved sensitivity. Am J Clin Pathol. 2007 Aug;128(2):282-6. doi: 10.1309/Q9W5HJTT24GQCXXX. PMID 17638663
- [Background] Aldous SJ, Richards M, Cullen L, Troughton R, Than M. Diagnostic and prognostic utility of early measurement with high-sensitivity troponin T assay in patients presenting with chest pain. CMAJ. 2012 Mar 20;184(5):E260-8. doi: 10.1503/cmaj.110773. Epub 2012 Jan 30. PMID 22291171
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284
- [Background] Hendel RC, Patel MR, Kramer CM, Poon M, Hendel RC, Carr JC, Gerstad NA, Gillam LD, Hodgson JM, Kim RJ, Kramer CM, Lesser JR, Martin ET, Messer JV, Redberg RF, Rubin GD, Rumsfeld JS, Taylor AJ, Weigold WG, Woodard PK, Brindis RG, Hendel RC, Douglas PS, Peterson ED, Wolk MJ, Allen JM, Patel MR; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American College of Radiology; Society of Cardiovascular Computed Tomography; Society for Cardiovascular Magnetic Resonance; American Society of Nuclear Cardiology; North American Society for Cardiac Imaging; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology. ACCF/ACR/SCCT/SCMR/ASNC/NASCI/SCAI/SIR 2006 appropriateness criteria for cardiac computed tomography and cardiac magnetic resonance imaging: a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group, American College of Radiology, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, American Society of Nuclear Cardiology, North American Society for Cardiac Imaging, Society for Cardiovascular Angiography and Interventions, and Society of Interventional Radiology. J Am Coll Cardiol. 2006 Oct 3;48(7):1475-97. doi: 10.1016/j.jacc.2006.07.003. No abstract available. PMID 17010819
- [Background] Hollander JE, Blomkalns AL, Brogan GX, Diercks DB, Field JM, Garvey JL, Gibler WB, Henry TD, Hoekstra JW, Holroyd BR, Hong Y, Kirk JD, O'Neil BJ, Jackson RE; Multidisciplinary Standardized Reporting Criteria Task Force. Standardized reporting guidelines for studies evaluating risk stratification of ED patients with potential acute coronary syndromes. Acad Emerg Med. 2004 Dec;11(12):1331-40. doi: 10.1197/j.aem.2004.08.033. No abstract available. PMID 15576525
- [Background] Bonaca M, Scirica B, Sabatine M, Dalby A, Spinar J, Murphy SA, Jarolim P, Braunwald E, Morrow DA. Prospective evaluation of the prognostic implications of improved assay performance with a sensitive assay for cardiac troponin I. J Am Coll Cardiol. 2010 May 11;55(19):2118-24. doi: 10.1016/j.jacc.2010.01.044. PMID 20447535
- [Background] Ronald J. Prineas RSC, Zhu-Ming Zhang. The minnesota code manual of electrocardiographic findings. London: Springer-Verlag; 2010.
- [Background] Rautaharju PM, MacInnis PJ, Warren JW, Wolf HK, Rykers PM, Calhoun HP. Methodology of ECG interpretation in the Dalhousie program; NOVACODE ECG classification procedures for clinical trials and population health surveys. Methods Inf Med. 1990 Sep;29(4):362-74. PMID 2233384
- [Background] Miller CD, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Mahler S, Diercks DB, Neiberg R, Hundley WG. Provider-directed imaging stress testing reduces health care expenditures in lower-risk chest pain patients presenting to the emergency department. Circ Cardiovasc Imaging. 2012 Jan;5(1):111-8. doi: 10.1161/CIRCIMAGING.111.965293. Epub 2011 Nov 29. PMID 22128195
- [Background] Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. Eur Heart J. 2000 Sep;21(18):1502-13. doi: 10.1053/euhj.2000.2305. PMID 10973764